CLINICAL TRIAL: NCT06478355
Title: Immunotherapy Combined With Chemoradiotherapy for First-line Treatment of Esophageal Squamous Cell Carcinoma:a Real-world Study From China
Brief Title: Immunotherapy Combined With Chemoradiotherapy for First-line Treatment of Esophageal Squamous Cell Carcinoma（ChinECR）
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024KY167
Record Dates: First submitted 2024-06-13; First posted 2024-06-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-06

CONDITIONS: ESCC
Keywords: ESCC; immunotherapy; chemoradiotherapy
MeSH Terms: interventions — Immunotherapy; Immune Checkpoint Inhibitors; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The patients with ESCC receive Immunotherapy combined with chemoradiotherapy (Experimental): Immunotherapy: intravenously, every 3 weeks for at least 6 months, or until progression, intolerance, or spontaneous withdrawal of the patient.
  Chemotherapy drug：albumin-bound paclitaxel 110-130mg/m2,d1,d8;cis-platinum 60-75mg/m2,d1 Q3W Radiotherapy: Total dose of 60Gy/30 times, each time 2.0Gy, 5 times a week from week 7 to week 12 of radiotherapy.
  Interventions: Drug: Immunotherapy; Drug: Chemotherapy drug; Radiation: radiotherapy

INTERVENTIONS:
Drug: Immunotherapy — Immunotherapy: intravenously, every 3 weeks for at least 6 months, or until progression, intolerance, or spontaneous withdrawal of the patient.
  Other Names: PD-1/PD-L1
Drug: Chemotherapy drug — TP:albumin-bound paclitaxel 110-130mg/m2,d1,d8;cis-platinum 60-75mg/m2,d1 Q3W
  Other Names: TP
Radiation: radiotherapy — Radiotherapy: Total dose of 60Gy/30 times, each time 2.0Gy, 5 times a week from week 7 to week 12 of radiotherapy.

SUMMARY:
This trial aims to assess efficacy and safety of immunotherapy combined with chemoradiotherapy for first-line treatment of esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Esophageal squamous cell carcinoma is a highly aggressive malignancy, with squamous cell carcinoma accounting for over 90% of esophageal cancer cases in China. According to the American Cancer Society, the 5-year survival rates vary among patients at different stages of esophageal cancer: approximately 50% for early and mid-stage cases, around 26% for locally advanced cases, and only 5% for those with distant metastasis.In recent years, immunotherapy combined with chemotherapy has emerged as the first-line standard treatment for advanced esophageal cancer, and several phase III trials of immunotherapy combined with radiotherapy are currently underway for locally advanced esophageal cancer. Despite being a novel treatment strategy for patients with locally advanced esophageal cancer, there remains a lack of sufficient evidence-based medical data supporting the use of immunotherapy combined with chemoradiotherapy.In recent years, immunotherapy combined with chemotherapy has emerged as the first-line standard treatment for advanced esophageal cancer, and several phase III trials of immunotherapy combined with radiotherapy are currently underway for locally advanced esophageal cancer. Despite being a novel treatment strategy for patients with locally advanced esophageal cancer, there remains a lack of sufficient evidence-based medical data supporting the use of immunotherapy combined with chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written signed informed consent;
* Age 18-85 years old, gender is not limited;
* Histologically or cytologically confirmed esophageal squamous cell carcinoma Exclusion Criteria,and patients with suspected brain or bone metastasis at the time of screening should undergo brain MRI or ECT before study enrollment;
* Physical status score ECOG 0-1;
* Weight > 40 kg;
* Expected survival ≥ 6 months;
* According to RECIST 1.1 guidelines, at least one lesion (not previously receiving radiotherapy) with a maximum diameter ≥ 10 mm as accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) at baseline (except lymph nodes, whose short axis must be ≥ 15 mm); And the lesion is suitable for repeated accurate measurement.;
* No previous immunotherapy;
* no serious abnormalities of haematopoietic, cardiac, pulmonary, hepatic; and renal functions and immunodeficiency (Haematology: white blood cells ≥3.5×109/L; neutrophils ≥1.5×109/L; haemoglobin ≥90g/L; platelets

  ≥100×109/L. Liver and kidney function: total bilirubin ≤1.5 times the upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) ≤2.5 times the upper limit of normal; creatinine ≤1.5 times the upper limit of normal; albumin ≥30 g/L. Coagulation: International Normalised Ratio (INR) or Prothrombin Time (PT) or Activated Partial Thromboplastin Time (APTT)

  ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, PT or INR is acceptable as long as the PT or INR is within the range of the anticoagulant drug formulation. Echocardiographic assessment: left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%). Pulmonary function FEV1 ≥70% of % of predicted value and DLCO ≥60% of % of predicted value).
* The female patient has evidence of postmenopausal status, or the urine or serum pregnancy test results of the premenopausal woman are negative. Women who stop menstruating for 12 months without other medical reasons are considered menopausal.

Exclusion Criteria:

* having any active autoimmune disease or a history of autoimmune disease (e.g. interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (which can be included if hormone replacement therapy is effective), etc.), and a history of immunosuppressive drug use within 28 days, with the exception of the use of hormones for the purpose of dealing with toxicity from radiotherapy;
* Previously received or are receiving other PD-1 antibody therapy or other immunotherapy targeting PD-1/PD-L1, or are currently participating in other interventional clinical studies for treatment;
* Have received other anti-tumour therapy (including herbal therapy with anti-tumour effect) within 4 weeks prior to the first dose of the study; have received long-term systemic immunotherapy or hormone therapy (except physiological replacement therapy, e.g., oral thyroxine for hypothyroidism) within 4 weeks prior to the first dose of the study; and have been treated with other experimental drugs or interventional clinical studies within 4 weeks prior to the first dose of the study;
* Patients with uncontrolled clinical cardiac symptoms or disease such as

  (1) NYHA class II or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
* with congenital or acquired immune function defects (e.g., HIV-infected patients), active hepatitis B (HBV-DNA ≥104 copies/ml) or hepatitis C (hepatitis C antibody-positive with HCV-RNA above the lower limit of detection of the analytical method), or active tuberculosis;
* Have an active infection or unexplained fever >38.5°C within 2 weeks prior to screening (at the investigator's discretion, subjects may be enrolled for fever arising from tumours);
* In the judgement of the investigator, the subject has other factors that may cause him/her to be forced to terminate the study in the middle of the study, e.g., suffering from other serious illnesses (including psychiatric illnesses) that require comorbid treatment, family or social factors that may affect the safety of the subject or the collection of trial data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of objective remission rate (ORR) in esophageal squamous cell carcinoma treated with immunotherapy combined with chemoradiotherapy | Treatment with immunotherapy for at least 6 months, or from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Objective remission rate (ORR): defined as the proportion of subjects whose tumor volume shrinks to a pre-specified value and can be maintained for the minimum time frame required, incorporating cases in complete remission (CR) and partial remission (PR).
Assessment of the incidence of treatment-related adverse events Incidence of Treatment-Emergent Adverse Events | Treatment with immunotherapy for at least 6 months, or from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Adverse events are observed during the course of the study and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE V5.0).

SECONDARY OUTCOMES:
Assessment of overall survival (OS) in esophageal squamous cell carcinoma | Treatment with immunotherapy for at least 6 months, or from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). OS is defined as the time from the start of enrollment to death from any cause.
Assessment of progression-free survival (PFS) in esophageal squamous cell carcinoma | Treatment with immunotherapy for at least 6 months, or from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). PFS is defined as the time from the start of enrollment until tumor progression or death from any cause.
Assessment of disease control rate (DCR) in esophageal squamous cell carcinoma | Treatment with immunotherapy for at least 6 months, or from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Disease control rate (DCR): the proportion of patients whose tumors shrank or were stable and remained so for a certain period of time, including complete remission (CR), partial remission (PR) and stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Shen, PhD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Liu X, Wen J, Zhang Y, Wang C, Liu Y, Qian P, Cao J, Hou Q, Xu Y, Lin Z, Ye X, Hou M, Gui Y, Wang L, Zhou W, Zeng Z, Song Y, Luo H, Lv J, Shen W. Impact of first-line chemoimmunotherapy with or without radiotherapy on the prognosis of patients with locally advanced or metastatic esophageal squamous cell carcinoma: a multicenter, real-world, retrospective cohort study from China (NCT06478355). Front Immunol. 2025 Jul 28;16:1633930. doi: 10.3389/fimmu.2025.1633930. eCollection 2025. PMID 40791599